CLINICAL TRIAL: NCT02018172
Title: Evaluation of the Adherence and the Patient Acceptability of Zomacton® Treatment With the Zomajet® Vision X Device
Acronym: ZOMAXEPT
Status: Terminated | Type: Observational
Why Stopped: Terminated due to lack of recruitment and difficulty in the selection of sites
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000122
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Growth Hormone Deficiency; Turner's Syndrome
MeSH Terms: conditions — Dwarfism, Pituitary; Turner Syndrome | interventions — Human Growth Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Zomacton® treatment with Zomajet® Vision X device
  Interventions: Drug: somatropin

INTERVENTIONS:
Drug: somatropin
  Other Names: Zomacton®

SUMMARY:
The study is performed to collect long-term data on the treatment adherence and patient's acceptability when Zomacton®10 mg is administered with the Zomajet® Vision X device in patients with a growth hormone deficiency or Turner's syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patient with growth hormone deficiency,

  1. Diagnosis of growth hormone deficiency proven by appropriate exploration
  2. Size ≤ -2 Standard Deviation (SD) according to the French references
  3. Growth velocity in the previous year inferior to the normal for age (-1SD) or < 4cm/year
* Growth deficiency due to Turner's syndrome

  1. Turner's syndrome confirmed by a karyotype
  2. Patient's size ≤ -2 SD according to the French references
  3. Bone age < 12 years
* Patient who require a minimum of 18 months of treatment.

Exclusion Criteria:

* There are no exclusion criteria except the contraindication for Zomacton® 10 mg

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a growth hormone deficiency or Turner's syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2014-07; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Rate of overall treatment adherence | Up to 18 months
  Ratio between actual duration of administration and total duration recommended by physician

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (1):
- Hôpital des Enfants, CHU de Toulouse, Toulouse, France